CLINICAL TRIAL: NCT00025285
Title: Phase II Study of Carboplatin, Irinotecan, and Thalidomide in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy Plus Thalidomide in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: REBACDR0000068946; CCCWFU-62400; NCI-5293
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Irinotecan; Thalidomide

INTERVENTIONS:
Drug: carboplatin
Drug: irinotecan hydrochloride
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining thalidomide with chemotherapy may kill more tumor cells and be an effective treatment for stage IIIB or stage IV non-small cell lung cancer.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus thalidomide in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and duration of response in patients with stage IIIB or IV non-small cell lung cancer treated with carboplatin, irinotecan, and thalidomide.
* Determine the progression-free and overall survival of patients treated with this regimen.
* Evaluate the toxicity profile of this regimen in these patients.

OUTLINE: Patients receive carboplatin IV over 30 minutes on day 1 and irinotecan IV over 90 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with stable or responsive disease receive up to 6 courses of therapy. Patients also receive oral thalidomide once daily beginning on day 1 and continuing until disease progression.

Patients are followed every 3 months until disease progression and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 39-70 patients will be accrued for this study within 14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IIIB (malignant pleural effusion) or stage IV non-small cell lung cancer

  * Squamous cell carcinoma
  * Basaloid carcinoma
  * Adenocarcinoma
  * Bronchoalveolar carcinoma
  * Adenosquamous carcinoma
  * Large cell carcinoma
  * Large cell neuroendocrine carcinoma
  * Giant cell carcinoma
  * Sarcomatoid carcinoma
  * Non-small cell carcinoma not otherwise specified
* Measurable disease

  * At least 1 unidimensionally measurable lesion

    * At least 20 mm by conventional techniques OR
    * At least 10 mm by spiral CT scan
  * The following lesions are considered nonmeasurable:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusions
    * Abdominal masses unconfirmed by imaging techniques
    * Cystic lesions
    * Previously irradiated brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception 4 weeks prior to, during, and for at least 4 weeks after thalidomide
* No prior seizures
* No other concurrent or prior malignancy within the past 5 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious medical or psychiatric illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except steroids for adrenal failure, hormones for non-cancer-related conditions (e.g., insulin for diabetes) or intermittent dexamethasone as an antiemetic

Radiotherapy:

* Prior radiotherapy for brain metastasis allowed if neurologically stable and off steroids
* No concurrent palliative radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-11-01 (Actual); Primary Completion 2004-09-29 (Actual); Study Completion 2004-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonius A. Miller, MD, Principal Investigator — Wake Forest University Health Sciences; James N. Atkins, MD, Principal Investigator — Southeastern Medical Oncology Center - Goldsboro
Locations (5):
- United States (5):
  - CCOP - Central Illinois, Decatur, Illinois
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina